CLINICAL TRIAL: NCT04054817
Title: A Multicenter, Open-label, Single-arm Study Assess the Collagen Ophthalmic Matrix for Anterior Lamellar Keratoplasty.
Brief Title: ACRO Biocornea Clinical Trial in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACRO Biomedical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-2017-01
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Corneal Ulcer
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Device: Lamellar keratoplasty-ABCcolla® Collagen Ophthalmic Matrix

INTERVENTIONS:
Device: Lamellar keratoplasty-ABCcolla® Collagen Ophthalmic Matrix — Lamellar keratoplasty was done by removing stromal layer, ABCcolla® Collagen Ophthalmic Matrix was sutured to the defective part of the cornea.
  Other Names: ACRO Biocornea

SUMMARY:
The goal of this clinical trial is to investigate the safety and clinical performance of ABCcolla Collagen Ophthalmic Matrix used for anterior lamellar keratoplasty in patients suffering from corneal ulcer.

Participants will undergo keratoplasty using the investigational product and be followed up for 24-week observation (total of 10 times).

ELIGIBILITY:
1. Inclusion criteria:

1. Male or female from 20 to 80 years old
2. Subject who has been diagnosed with corneal ulcer
3. The depth or the size of the ulcer increases or increased anterior chamber inflammation after treatment (clinic, hospitalization, or others…)
4. The corneal ulcer affects corneal stroma depth to 1/3 and infiltrates >2 mm diameter, detected by OCT
5. Best corrected vision acuity < 0.05
6. Subject who signs the informed consent form (ICF), and agrees to complete the treatment and follow-up

2. Exclusion criteria:

1. Accepted keratoplasty
2. Has a corneal perforation and expects to have vision
3. Has a severe dry eye
4. Experience s incomplete eyelid closure
5. H as liver function (ALT and AST) tests with the score as twofold or greater than that of the normal
6. Has renal function (Cr) levels greater than normal two folders
7. Has serum protein 10% low than normal
8. Has severe cardiovascular and cerebral vascular disease
9. Subject with uncontrolled diabetes
10. Subject with current malignancy
11. Known to be allergic to collagen
12. Has a systemic collagen connective tissue disease
13. Has a constitution prone to severe allergic reactions
14. Use s anticoagulants 5 days before studying keratoplasty
15. Use s injectable NSAID 3 days before studying keratoplasty
16. Cannot accept investigated material due to religious or cultural reason
17. Pregnant or breastfeeding women or childbearing-age women who plan to get pregnant
18. Participation in any drug or medical device clinical trial within 30 days prior to signing the informed consent form;
19. Not being considered suitable for this study by the investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Incidence rate of irreversible graft dissociation or irreversible graft rejection within 6 months. | After the surgery, patients will be examined for follow-up observation for 24 weeks.
  Count the number of subjects with irreversible graft dissolution or irreversible rejection within 24 weeks, and calculate the incidence rate

SECONDARY OUTCOMES:
The extent of graft transparency | 24-week follow-up visit. Totoa 9 times.
  After examined via slit lamp by the clinical ophthalmologist, the graft transparency were graded from 0 to 4, which indicated transparency, slight turbidity, mild turbidity of matrix and visble iris, worsening turbidity with invisible iris, and invisible pupil, respectively.
The extent of graft vascularization | 24-week follow-up visit. Totoa 9 times.
  After examined via slit lamp by the clinical ophthalmologist, the extent of neovascularization was grades 0 if there were none, 1-4 if neovascularization had grown into the corneal limbus, the border of graft, 2mm of the gtaft, and into the center of the graft, respectively.
Infection recurrence | 24-week follow-up visit. Totoa 9 times.
  The recurrence was examined via slit lamp by the clinical ophthalmologist.
The extend of corneal edema | 24-week follow-up visit. Totoa 9 times.
  After examined via OCT by the clinical ophthalmologist, the corneal edema were graded from none, mild, moderate and severe by the doctor.
Best corrected vision acuity | 24-week follow-up visit. Totoa 9 times.
  Examied by the Optometer.
Light sensitivity | 24-week follow-up visit. Totoa 9 times.
  The light perception was tested by the clinical ophthalmologist.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Cheng Tai, MD, Principal Investigator — Tri-Service General Hospital
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang YH, Tseng FW, Chang WH, Peng IC, Hsieh DJ, Wu SW, Yeh ML. Preparation of acellular scaffold for corneal tissue engineering by supercritical carbon dioxide extraction technology. Acta Biomater. 2017 Aug;58:238-243. doi: 10.1016/j.actbio.2017.05.060. Epub 2017 Jun 1. PMID 28579539